CLINICAL TRIAL: NCT04251091
Title: Ankle Exosuit Training in the Clinic to Community
Brief Title: Ankle Exosuit Training in the Clinic to Community Community
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arun Jayaraman, PT, PhD (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Organization: Shirley Ryan AbilityLab (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00209869
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: exoskeleton; ambulation; robotics; Stroke; walking
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Previous work has demonstrated that the tuning of the exosuit technology is important for each patient post stroke to be able to maximally utilize the technology. These modulations include when the plantarflexion force is delivered, and how to deliver the assistance within a training session however it is still unclear how to implement this into a training protocol. During a part of this study, we will explore which timing: early timing (10-20%), mid timing (50%) and late timing (90%) may be optimal for an individual and then carry out a training protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReWalk Soft Exosuit (Experimental): During this study, we will explore which timing: early timing (10-20%), mid timing (50%) and late timing (90%) may be optimal for an individual and then carry out an 18 session training protocol.
  Interventions: Other: Treadmill walking; Other: Overground Walking

INTERVENTIONS:
Other: Treadmill walking — Up to 5 bouts of 6 minutes walking on the treadmill with rest breaks allowed between sets
Other: Overground Walking — Up to 5 bouts of 6 minutes walking overground with rest breaks allowed between sets

SUMMARY:
This study focuses on investigating exosuit technology by evaluating its ability to provide a gait-restorative effect delivered in both clinic and community settings. The exosuit provides dynamic dorsiflexion and plantarflexion assist during walking. We will determine the effect of training parameters of intensity, repetition, and gait quality which are all key parameters associated with experience-dependent neuroplasticity. The other objective is to determine the effect of this intervention on community walking activity, walking speed, walking distance, and locomotor mechanics and energetics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years old
* Stroke event occurred at least 6 months ago
* Observable gait deficits
* Able to walk without the support of another person for at least 2 minutes (with or without an assistive device or orthotic support)
* Passive ankle dorsiflexion range of motion to neutral with the knee extended (i.e., able to achieve an angle of 90 degrees between the shank and the foot)
* Resting heart rate between 40 - 100 bpm, inclusive
* Resting blood pressure between 90/60 and 170/90 mmHg, inclusive
* Medical clearance by a physician

Exclusion Criteria:

* Score of >1 on question 1b and >0 on question 1c on the NIH Stroke Scale
* Inability to communicate with investigators
* Neglect or hemianopia
* Unexplained dizziness in the last 6 months
* Pressure ulcers or skin wounds located at human-device interface sites
* History of significant Peripheral Artery Disease (PAD)
* Unresolved Deep Vein Thrombosis (DVT)
* Uncontrolled or untreated hypertension
* Significant paretic ankle contractures (plantarflexion > 5°)
* Psychiatric or cognitive impairments that may interfere with proper operation of the device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 10 Meter Walk Test from baseline gait speed | Baseline Day 1-3, Midpoint at week 6, Post-intervention at week 12
  This test will examine the patient's gait speed. Patients will be directed to walk at their preferred and maximum but safe speed. Patients will be positioned 1 meter before the start line and instructed to walk the entire distance and past the end line approximately 1 meter. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundredth of a second (ex: 2.15 sec).

SECONDARY OUTCOMES:
Change in 6 Minute Walk Test in distance from baseline | Baseline Day 1-3, Midpoint at week 6, Post-intervention at week 12
  The 6 Minute Walk Test (6MWT) measures the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The test will be used to determine participant's gait efficiency at baseline and at study completion. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded.
Functional Gait Assessment (FGA) | Baseline Day 1-3, Midpoint at week 6, Post-intervention at week 12
  The Functional Gait Assessment is a 10 item test used to assess postural stability during walking tasks. It has a maximum score of 30 with each item being scored 0-3. It may be performed with or without an assistive device; however, individuals lose a point on all items requiring a device.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

REFERENCES:
- [Derived] Shin SY, Hohl K, Giffhorn M, Awad LN, Walsh CJ, Jayaraman A. Soft robotic exosuit augmented high intensity gait training on stroke survivors: a pilot study. J Neuroeng Rehabil. 2022 Jun 3;19(1):51. doi: 10.1186/s12984-022-01034-2. PMID 35655180